CLINICAL TRIAL: NCT04277403
Title: Hippocampal Avoidance Whole Brain Radiotherapy (HA-WBRT) and Stereotactic Radiosurgery (SRS) in Patients With Multiple Brain Metastases
Brief Title: HA-WBRT vs SRS in Patients With Multiple Brain Metastases
Acronym: HipSter
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIPSTER_2020
Record Dates: First submitted 2020-02-06; First posted 2020-02-20 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Brain Metastases
Keywords: brain metastases; hippocampal avoidance; radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Observer-blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA-WBRT+SIB (Experimental): Hippocampal avoiding Whole brain radiation therapy (HA-WBRT) with volumetric modulated arc therapy (VMAT) with a simultaneously integrated boost (SIB) to each brain metastasis
  Interventions: Radiation: Hippocampal Avoiding Whole Brain Radiation Therapy with Simultaneous Integrated Boost
- SRS (Active Comparator): Single session or hypofractionated stereotactic radiosurgery (SRS) of multiple brain metastases
  Interventions: Radiation: Single session or hypofractionated stereotactic radiosurgery

INTERVENTIONS:
Radiation: Hippocampal Avoiding Whole Brain Radiation Therapy with Simultaneous Integrated Boost — Hippocampal avoiding Whole brain radiation therapy (HA-WBRT) with volumetric modulated arc therapy (VMAT) with a prescribed dose of 30Gy in 12 fractions, 2.5Gy per fraction and a simultaneously integrated boost (SIB) to each brain metastasis of 51Gy to 95% of PTV in 12 Fractions, 4.25Gy per fraction.
  Arms: HA-WBRT+SIB
Radiation: Single session or hypofractionated stereotactic radiosurgery — Single session or hypofractionated stereotactic radiosurgery (SRS) of multiple brain metastases. Single session SRS will be delivered in 18 to 22Gy to the tumour encompassing 80% Isodose. Hypofractionated stereotactic radiosurgery (HfSRS) will be delivered in 5 sessions of 6Gy each to the tumour encompassing 80% isodose.
  Arms: SRS

SUMMARY:
This study compares the effectiveness and safety of two radiation treatment techniques for patients with multiple brain metastases.

DETAILED DESCRIPTION:
For patients suffering from multiple brain metastases whole brain radiation therapy still constitutes a standard therapy. However, because of the risk of neurocognitive side effects as well as reduced local tumor control, employment of stereotactic radiosurgery (SRS) is becoming more common. The disadvantage of SRS alone may be poor intracranial tumor control because of frequent appearance of new distant brain metastases after therapy. In recent years hippocampal avoidance whole brain therapy has been shown to minimize treatment related side effects while reducing the rate of distant intracranial failure.

In this study patients will be randomized to receive either hippocampal avoidance whole brain radiation therapy with integrated tumor boost (HA-WBRT+SIB) or stereotactic radiosurgery. The investigators hypothesize that HA-WBRT+SIB can improve intracranial tumor control compared to stereotactic radiosurgery, while avoiding additional neurocognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 and not exceeding 15 brain metastases not exceeding a combined total volume of 25ml and not previously treated with radiotherapy
* KPI ≥ 70, ECOG ≤ 2
* Age ≥ 18 years, Male or female

Exclusion Criteria:

* Neuroendocrine, SCLC, germinoma or lymphoma histology
* Brain stem metastasis
* Life expectancy < 3 months
* Suspicion of meningeosis carcinomatosa
* Previous WBRT
* Inability to participate in radiologic follow-up, contraindication to MR imaging (e.g. not MRI compatible pacemaker, severe claustrophobia)
* Inability to participate in neurocognitive function testing, insufficient German language skills, aphasia, graphomotor impairment, insufficient vision, insufficient attention span
* Pregnancy, nursing or unwillingness to prevent pregnancy using effective methods of contraception during treatment
* Known abuse of medication, drugs or alcohol
* Known severe dementia (z-score < 2) or major cognitive function disorder that is not caused by intracranial tumour
* Known clinical depression or psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progression free survival | up to 18 months
  survival with freedom from both local and distant intracranial progression, measured in months from end of treatment until progression or death, assessed in follow-up imaging (MRI, FET-PET)

SECONDARY OUTCOMES:
Neurocognitive function assessed by VLMT | up to 18 months
  Change of z-scores of VLMT (Verbaler Lern- und Merkfähigkeitstest) to baseline examination
Neurocognitive function assessed by COWAT | up to 18 months
  Change of z-scores of COWAT (controlled oral word association test) to baseline examination
Neurocognitive function assessed by TMT | up to 18 months
  Change of z-scores of TMT (trail making test) to baseline examination
Local control rate | up to 18 months
  rate of progression of treated metastases assessed in follow-up imaging (MRI, FET-PET)
Survival time | up to 18 months
  time from end of treatment to death
Quality of Life Score assessed by EORTC QLQ-C30 questionnaire | up to 18 months
  Change in Quality of Life Score of EORTC QLQ-C30 (Quality of life core module) relative to baseline
Quality of Life Score assessed by QLQ-BN20 questionnaire | up to 18 months
  Change in Quality of Life Score of QLQ-BN20 (quality of life brain cancer module) relative to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Undecided